CLINICAL TRIAL: NCT03310424
Title: Transcriptomic and Next Generation Sequencing Approaches to Infection With Treponema Pallidum
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 14423
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Lesion Swab samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No active intervention. — No active intervention is undertaken. Collection of samples for bio-informatic analysis only

SUMMARY:
Syphilis is an important sexually transmitted infection. There has been an epidemic of syphilis amongst men who have sex with men in the United Kingdom in the last decade. Early infection with syphilis causes a genital ulcer followed, in the absence of treatment, by a generalised illness often accompanied by rash. Studies on the pathogenesis of syphilis have been limited because it is not possible to grow syphilis outside of the body. New approaches using molecular tests allow the immune response of the patient to infection to be measured directly from a swab of a genital ulcer or rash and/or a blood sample and also allow the whole genetic sequence of the bacteria to be obtained from a swab.

In this study the investigators will collect swabs from ulcers or rashes and a blood sample from patients with syphilis and measure both the response of the patient immune system and the genetic sequence of the bacteria. Patients will be enrolled at sexual health clinics in the United Kingdom. Patients will receive standard medical care including standard treatment for syphilis in line with national guidelines. Standard management already includes collection of a swab and a blood sample. For this study an additional swab sample and an additional 5ml of blood will be collected for use in this research project. By better understanding host immune system responds to infection with syphilis the studies aims to gain better insights in to the pathogenesis of this important sexually transmitted disease.

ELIGIBILITY:
Inclusion Criteria:

* Early infectious syphilis with exudative skin/genital lesions from which a lesion swab can be obtained

Exclusion Criteria:

* Age <18 years
* Unable to provide consent
* Patients with other stages of syphilis apart from Primary or Secondary OR patients without a lesion from which swabs can be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early infectious syphilis with exudative skin/genital lesions from which a lesion swab can be obtained
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Whole Genome Sequencing | From samples collected at baseline
  Whole Genome Sequencing of T.pallidum
Host Transcriptomic Response | From samples collected at baseline
  RNA Sequencing from lesion and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Mortimer Market Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes